CLINICAL TRIAL: NCT00366509
Title: Role of Helicobacter Pylori and Its Toxins in Pulmonary and Oropharyngeal Disease
Brief Title: Role of Helicobacter Pylori and Its Toxins in Lung and Digestive System Diseases
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060222; 06-H-0222
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Disease; Oropharyngeal Disease; Lymphangioleiomyomatosis; Pulmonary Fibrosis; Asthma; Sarcoidosis
Keywords: Vac A Toxin; Lung; Bronchoscopy; Endoscopy; Cytotoxin; Pulmonary Disease; Lung Disease; Genetic Disease; Oropharyngeal Disease; Pulmonary Fibrosis; Asthma
MeSH Terms: conditions — Lung Diseases; Lymphangioleiomyomatosis; Pulmonary Fibrosis; Asthma; Sarcoidosis; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Lung Disease
- 2: Healthy volunteer

SUMMARY:
This study will examine bacteria and toxins in the mouth, lung and digestive system that may be the cause of various diseases or symptoms. H. pylori is a bacterium that produces various toxins that may contribute to lung problems. This study will examine specimens collected from the mouth, teeth, lung, digestive tract and blood to measure H. pylori and its toxins and their effects on cells.

People 18 years of age and older with or without gastrointestinal disease may be eligible for this study. These include people without a history of lung disease as well as patients with any of the following: lymphangioleiomyomatosis, asthma, sarcoidosis, other chronic or genetic lung disease (e.g., chronic obstructive pulmonary disease, cystic fibrosis or eosinophilic granuloma).

Participants may undergo the following tests:

* Blood and urine tests, chest x-ray.
* Measurement of arterial blood gases: A small needle is placed in an artery in the forearm to collect arterial blood.
* Lung function tests: Subjects breathe deeply and occasionally hold their breath. They may also receive a medication that expands the airways.
* Fiberoptic bronchoscopy with lavage and bronchial brushing: The subject's mouth and throat are numbed with lidocaine; a sedative may be given for comfort. A thin flexible tube called a bronchoscope is advanced through the nose or mouth into the lung airways to examine the airways. Saline (salt water) is then injected through the bronchoscope into the air passage and then removed by gentle suction. Next, a small brush is passed through the bronchoscope and an area of the airway is brushed to collect some cells for examination.
* Mouth rinsing or teeth brushing to collect cells.
* Endoscopy: A small needle and catheter (thin plastic tube) are placed into an arm vein to administer fluids and medications through the vein. A sedative may be given. The throat is numbed with lidocaine and a thin flexible tube called an endoscope is inserted through the mouth and down the esophagus into the stomach and upper part of the small intestine to examine those areas.

DETAILED DESCRIPTION:
Vacuolating cytotoxin A (VacA toxin), an 88-kDa multifunctional protein, and other toxins are produced by Helicobacter pylori. We hypothesize that H. pylori, VacA toxin, and other toxins within the gastrointestinal tract and/or oropharynx are also found in the lung and may contribute to decline in lung function. Analyses of gastrointestinal, oropharyngeal, lung and blood specimens will improve the understanding of H. pylori, VacA toxin, and other toxins as well as their potential role in pathophysiology of disease. The objectives of this exploratory protocol are to procure gastrointestinal, oropharyngeal, lung and/or blood specimens from healthy research volunteers and subjects with lung disease (e.g., lymphangioleiomyomatosis, asthma, sarcoidosis, pulmonary fibrosis) and to analyze these specimens for H. pylori, VacA toxin, and other toxins. We hypothesize that the toxins may have a role in the pathogenesis of lung disease and in the subclinical decline in lung function seen with aging.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals who are 18 years of age or older with or without a history of gastrointestinal disease and with any of the following:

1. lymphangioleiomyomatosis, or
2. asthma, or
3. sarcoidosis, or
4. pulmonary fibrosis, or
5. other chronic or genetic lung diseases (e.g., chronic obstructive pulmonary disease, eosinophilic granuloma, cystic fibrosis, Wegener's granulomatosis, chronic bronchitis), or
6. research volunteers without a history of lung disease.

EXCLUSION CRITERIA:

Individuals with any of the following:

1. uncontrolled ischemic heart disease, or
2. uncorrectable bleeding diathesis, or
3. pregnancy or lactation, or
4. inability to give informed consent, or
5. risk factors for endocarditis (e.g., prosthetic cardiac valve, previous bacterial endocarditis, surgically constructed systemic pulmonary shunts or conduits, complex cyanotic congenital heart disease [e.g., single ventricle, transposition of great arteries, tetralogy of Fallot])

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 139 patient volunteers and 18 healthy research volunteers have participated in this protocol at the NIH. 133 female patients with lymphangioleiomyomatosis (age range at accrual from 22 to 72 years old: 121 white, 7 black, 4 asian, and 1 unknown). 2 female patients with other chronic/genetic lung diseases (age range at accrual from 47 to 71: 2 white). 4 male patients with pulmonary fibrosis (age range at accrual from 67 to 74: 4 white). 18 research volunteers without lung disease (age range at accrual from 19 to 67: 6 white males, 5 white females, 5 black females, 1 hispanic multi-race male, and 1 hispanic unknown male.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2006-09-18 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-10-27 (Actual)

PRIMARY OUTCOMES:
procure and analyze gastrointestinal, oropharyngeal, lung and/or blood specimens from healthy research volunteers and subjects with lung disease | ongoing
  Procure and analyze gastrointestinal, oropharyngeal, lung and/or blood specimens from healthy research volunteers and subjects with lung disease (e. g., lymphangioleiomyomatosis, asthma, sarcoidosis, pulmonary fibrosis). Comparison of specimens from subjects may further the understanding of H. pylori, VacA cytotoxin, and/or other toxins in oropharyngeal, pulmonary, and gastrointestinal conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cover TL, Blanke SR. Helicobacter pylori VacA, a paradigm for toxin multifunctionality. Nat Rev Microbiol. 2005 Apr;3(4):320-32. doi: 10.1038/nrmicro1095. PMID 15759043
- [Background] Hocker M, Hohenberger P. Helicobacter pylori virulence factors--one part of a big picture. Lancet. 2003 Oct 11;362(9391):1231-3. doi: 10.1016/S0140-6736(03)14547-3. PMID 14568748
- [Background] Israel DA, Peek RM. pathogenesis of Helicobacter pylori-induced gastric inflammation. Aliment Pharmacol Ther. 2001 Sep;15(9):1271-90. doi: 10.1046/j.1365-2036.2001.01052.x. PMID 11552897
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-H-0222.html